CLINICAL TRIAL: NCT04832932
Title: A Phenotypic Study of Safety, Tolerability, Reactogenicity, Immunogenicity, and Virus Shedding With Post-Vaccination Infections of Emergency-Use-Authorized Vaccines Against COVID-19
Brief Title: The COVID-19 Back-to-Normal Study: Analysis of Multiple Outcomes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mebo Research, Inc. (Other)
Collaborators: Aurametrix (Other)
Responsible Party: Sponsor
Other Study IDs: 20210103MEBO
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: COVID-19 Vaccines
Keywords: Drug-Related Side Effects and Adverse Reactions; Long-term adverse effects; Immunogenicity, Vaccine; COVID-19
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Long Term Adverse Effects; COVID-19 | interventions — COVID-19 Vaccines; BNT162 Vaccine; 2019-nCoV Vaccine mRNA-1273; Ad26COVS1; ChAdOx1 nCoV-19; sinovac COVID-19 vaccine; BIBP COVID-19 vaccine; BBV152 COVID-19 vaccine; NVX-CoV2373 adjuvated lipid nanoparticle

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (6):
- 80 years of age or older: Individuals 80-89, 90-99, 100 years of age and older who received COVID-19 vaccine
  Interventions: Biological: COVID-19 vaccines
- 60-79 years of age: Individuals 60-69 and 70-79 years of age who received COVID-19 vaccine
  Interventions: Biological: COVID-19 vaccines
- 40-59 years of age: Individuals in 40-49, 50-59 age range who received COVID-19 vaccine
  Interventions: Biological: COVID-19 vaccines
- 18-39 years of age: Individuals in 18-29, 30-39 age range who received COVID-19 vaccine
  Interventions: Biological: COVID-19 vaccines
- MEBO/PATM: Individuals with present or past MEBO/PATM symptoms who received COVID-19 vaccine
  Interventions: Biological: COVID-19 vaccines
- Chronic Disease: Individuals with self-reported chronic health conditions who received COVID-19 vaccine
  Interventions: Biological: COVID-19 vaccines

INTERVENTIONS:
Biological: COVID-19 vaccines — Emergency-use authorized COVID-19 vaccines
  Other Names: BNT162b2; mRNA-1273; JNJ-78436735; AZD1222; Gam-KOVID-Vak; CoronaVac/Sinovac; BBIBP-CorV; BBV152; NVX-CoV2373

SUMMARY:
During the study, members of different online and offline communities will be followed post COVID-19 vaccination.

Injection-site (local) and systemic reaction data will be assessed on vaccination day and afterwards using either web surveys or personal communication, depending on study participant preference.

Hypothesis to be tested: The safety profile and the magnitude and durability of immune responses to the COVID-19 vaccines as well as adverse reactions depend on health conditions, metabolism and microbiomes.

DETAILED DESCRIPTION:
The outbreak of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) was declared a Public Health Emergency of International Concern in January 2020 and upgraded to pandemic in March 2020. First vaccines to prevent COVID-19 were authorized for emergency use in the US in December 2020, but a number of unknowns still remains. One of these unknowns is the relationship of the microbiota, gut dysbiosis and impaired metabolism with active immunity to pathogens and vaccines and tolerance to antigens. Study groups will be based on age, metabolism, donated diagnostic test results and self-reported symptoms. Data will be collected continuously via surveys and investigator-participant interactions, as needed. Statistical methods used will be the ones with the greatest power.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 or older at the time of consent
* Intention to vaccinate and of being available for entire study period

Exclusion Criteria:

* Any illness or condition that in the opinion of the investigator may affect the safety of the participant or the evaluation of any study endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals 18 or older interested in vaccinating
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2025-01-05 (Estimated)

PRIMARY OUTCOMES:
Adverse reactions/events | 10 days after any dose of study intervention.
  Percentage of occurrence, types, duration and severity of adverse events occurring within 10 days post-doses 1 and 2

SECONDARY OUTCOMES:
Long-term adverse events | Throughout the study period, until 12 months post-final-dose
  Percentage of occurrence, types, duration and severity of adverse events throughout study period
Incidence of COVID-19 cases | From 14 days after completion of the 2-dose regimen up to 12 months post-final-dose
  The number of COVID-19 cases occurring <=14 or ≥ 15 days after any dose of study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Gabashvili, PhD, Principal Investigator — Mebo Research, Inc.
Locations (5):
- United States (2):
  - MEBO Research, Inc, Miami, Florida
  - Kahite, Vonore, Tennessee
- Gabashvili, Tbilisi, Georgia
- MEBO Research Africa, Kilifi, Kenya
- Mebo Research (Uk), London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No
individual participant data will remain confidential, unless specifically requested to be shared by the participant

REFERENCES:
- [Result] Gabashvili IS. The Incidence and Effect of Adverse Events Due to COVID-19 Vaccines on Breakthrough Infections: Decentralized Observational Study With Underrepresented Groups. JMIR Form Res. 2022 Nov 4;6(11):e41914. doi: 10.2196/41914. PMID 36309347
- See also: Study updates — https://www.aurametrix.com/nct04832932.html